CLINICAL TRIAL: NCT05146791
Title: Clinical and Radiographic Outcomes in Arthroscopic Cuistow Procedure and Arthroscopic Modified Bristow Procedure
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021039-2
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Shoulder Dislocation
Keywords: Bristow; shoulder dislocation; Inlay
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inlay Bristow Group: Inlay Bristow procedure
  Interventions: Procedure: Inlay Bristow
- Onlay Bristow Group: Onlay Bristow procedure
  Interventions: Procedure: Bristow

INTERVENTIONS:
Procedure: Inlay Bristow — A modified Bristow procedure
  Other Names: Cuistow
  Groups: Inlay Bristow Group
Procedure: Bristow — Traditional Bristow procedure
  Other Names: Modified Bristow procedure
  Groups: Onlay Bristow Group

SUMMARY:
To evaluate the clinical and radiographic outcomes of arthroscopic Chinese Unique Inlay Bristow procedure (Cuistow procedure) and arthroscopic Bristow procedure in treating recurrent anterior shoulder instability.

DETAILED DESCRIPTION:
Aim: To compare the clinical and radiographic outcomes following the arthroscopic Chinese Unique Inlay Bristow (Cuistow) procedure and the arthroscopic Bristow procedure.

Background: The Cuistow procedure is a modified Bristow surgery in which a Mortise and Tenon structure was added to the contact surface between the coracoid tip and the glenoid. In previous study, patients received Cuistow procedure have satisfying clinical performance and excellent postoperative bone healing rate (96.1%). However, no comparative studies was performed.

Study Design: Retrospective comparative case-cohort study

Methods: Patients who underwent the arthroscopic Cuisotw procedure and modified Bristow procedure between Jan 2017 and Mar 2018 were selected. 70 patients with recurrent anterior shoulder instability were included. Radiological evaluations with 3D CT scan were performed preoperatively, immediately after the operation, and postoperatively at three months and during the final follow-up (more than 2 years). Clinical assessment for a minimum of 24 months including the 10-point visual analog scale for pain and subjective instability, University of California at Los Angeles scoring system (UCLA score), American Shoulder and Elbow Surgeons score (ASES score), ROWE score, Subjective Shoulder Value (SSV) and active range of motion were completed by independent observers and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. a glenoid defect ≥10% but <25%,
2. participation in high-demand (collision and overhead) sports combined with the presence of a glenoid defect <25% of the glenoid or without defect
3. failure after Bankart repair.

Exclusion Criteria:

1. multidirectional shoulder instability (MDI),
2. uncontrolled epilepsy
3. pathological involvement of other soft tissue such as the long head of the biceps or a rotator cuff tear
4. previous shoulder stability surgery other than Bankart repair
5. Follow-up was less than 2 years or incomplete follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients undergoing the Cuistow procedure and modified Bristow procedure in our hospital between Jan 2017 and Mar 2018.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Bone union rate | 3-month postoperatily
  Bone healing was observed in 3D-CT. The bone healing rate was obtained by dividing the number of people who achieved bone healing by the total number of people.
Bone union rate | 2-year postoperatily
  Bone healing was observed in 3D-CT. The bone healing rate was obtained by dividing the number of people who achieved bone healing by the total number of people.
ASES score | 2-year postoperatively
  The ASES score (Michener 2002) is a 10-item measure of shoulder pain and function. Pain is assessed on a 10-cm visual analog scale (VAS) and accounts for 50% of the total score. The remaining 50% of the score is determined by the responses to 10 4-point Likert-scale questions related to physical function.

SECONDARY OUTCOMES:
dislocation rate | 2-year postoperatively
  The dislocation rate was obtained by dividing the number of people who dislocated postopratively by the total number of people.
VAS for pain score | 2-year postoperatively
  The visual analog scale (VAS) for pain score is the most commonly used to describe pain levels in patients, ranging from 0 to 10, with a higher score indicating more intense pain.
Active shoulder ranges of motion | 2-year postoperatively
  internal rotation at the side, and external and internal rotation at 90° of abduction

CONTACTS AND LOCATIONS:
Locations (1):
- PekingUTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No